CLINICAL TRIAL: NCT00021138
Title: Computerized Scheduling of Nicotine Inhaler Use
Brief Title: Computer-Assisted Scheduling of Nicotine Inhaler Use in Participants Who Plan to Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Personal Improvement Computer Systems (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: PICS-R44-CA80525; CDR0000068751 (Registry Identifier: PDQ (Physician Data Query)); NCI-V01-1662
Record Dates: First submitted 2001-07-11; First posted 2004-03-19 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2011-03

CONDITIONS: Esophageal Cancer; Head and Neck Cancer; Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer; esophageal cancer; hypopharyngeal cancer; laryngeal cancer; nasopharyngeal cancer; oropharyngeal cancer; lip and oral cavity cancer; paranasal sinus and nasal cavity cancer; tongue cancer
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Mouth Neoplasms; Tongue Neoplasms | interventions — Nicotine

INTERVENTIONS:
Behavioral: smoking cessation intervention
Drug: nicotine

SUMMARY:
RATIONALE: Computer-assisted scheduling of nicotine inhaler use may be an effective method to help people stop smoking.

PURPOSE: Randomized cinical trial to compare the effectiveness of computer-assisted scheduling of nicotine inhaler use with that of self-scheduled nicotine inhaler use in participants who plan to stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of program length on inhaler use compliance, latency to smoking relapse, and gradual cessation of inhaler use in participants using a computer-assisted program to schedule nicotine inhaler dosing for smoking cessation. II. Compare fast and slow paced versions of computer-assisted scheduling of nicotine inhaler use versus ad libitum nicotine inhaler use, in terms of smoking cessation rates, in these participants. III. Compare these dosing conditions, in terms of adherence, initial dosing levels, and successful tapering effects, in these participants.

OUTLINE: This is a randomized study. Participants are randomized to one of three arms. All participants monitor their period of cigarette smoking for 7 days by pressing a data input button on a hand-held computer every time they smoke. Arm I: Participants begin using a nicotine inhaler according to the dosing instructions that come with it and monitor their inhaler usage with the hand-held computer. Arm II: Participants are prompted by the hand-held computer to use a nicotine inhaler based on their prior smoking habits. When prompted, participants use the nicotine inhaler at a comfortable rate over 20 minutes. The computer prompts participants at a fixed frequency and duration of inhaler use for 3 weeks and then tapers the frequency and duration over 3-5 weeks. Arm III: Participants are prompted by the hand-held computer and use a nicotine inhaler as in arm II. The computer prompts participants at a fixed frequency and duration of inhaler use for 12 weeks and then tapers the frequency and duration over 3-5 weeks. Participants keep a weekly diary of the average number of cigarettes smoked, average number of inhaler sessions, and average length of each session. Participants also record the date of any 24-hour smoking cessation and relapse and complete a withdrawal symptoms questionnaire. Participants are followed at 1 year.

PROJECTED ACCRUAL: A total of 480 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Smoker with a daily smoking rate between 15 and 40 cigarettes per day for at least 2 years Willing to quit smoking Willing to use a nicotine inhaler No concurrent use of smokeless tobacco, pipes, or cigars

PATIENT CHARACTERISTICS: Age: 18 to 67 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No liver disease Renal: No kidney disease Cardiovascular: No history of heart disease No high blood pressure Other: No stomach ulcers No overactive thyroid Not pregnant or nursing No plans to become pregnant within the next 6 months

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No concurrent insulin Radiotherapy: Not specified Surgery: Not specified Other: At least 1 month since prior bupropion or antidepressants At least 1 year since prior treatment for substance abuse No other concurrent nicotine replacement products

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Riley, PhD, Study Chair — Personal Improvement Computer Systems
Locations (1):
- Personal Improvement Computer Systems, Incorporated, Reston, Virginia, United States